CLINICAL TRIAL: NCT05250193
Title: A Prospective, Multi-center, Randomized Study to Evaluate the Safety and Efficacy of DK ScoreTM Scoring Balloon Vesus Non-Slip Element Coronary Dilatation Catheter for Coronary Artery Stenosis
Brief Title: DK Score Coronary Scoring Balloon: a RCT Trial to Evaluate Acute Lumen Gain (SCORE CHINA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DK Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-P-2019-006
Record Dates: First submitted 2022-02-05; First posted 2022-02-22 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Coronary Stenosis
Keywords: Scoring balloon; DK Score; NSE
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DK ScoreTM Coronary Scoring Balloon (DK Score) (Experimental): DK ScoreTM Coronary Scoring Balloon Manufactured by DK Medical Technolgy CO.,LTD
  Interventions: Device: DK ScoreTM Coronary Scoring Balloon
- Non-Slip Element Coronary Dilatation Catheter (NSE) (Active Comparator): Non-Slip Element Coronary Dilatation Catheter Manufactured by GOODMAN CO.,LTD
  Interventions: Device: Non-Slip Element Coronary Dilatation Catheter

INTERVENTIONS:
Device: DK ScoreTM Coronary Scoring Balloon — After pre-dilation balloon is used (if any), DK Score is used as final dilatation balloon before Drug Eluting Stent implantation or Drug Coated Balloon deployment.
  Other Names: DK Score
  Arms: DK ScoreTM Coronary Scoring Balloon (DK Score)
Device: Non-Slip Element Coronary Dilatation Catheter — After pre-dilation balloon is used (if any), NSE is used as final dilatation balloon before Drug Eluting Stent implantation or Drug Coated Balloon deployment.
  Other Names: NSE
  Arms: Non-Slip Element Coronary Dilatation Catheter (NSE)

SUMMARY:
A prospective, Multi-center, Randomized Study designed to evaluate the acute lumen gain and device procedural success of the DK ScoreTM Scoring balloon versus NSE Scoring Balloon for patients with coronary arteries stenosis.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized controlled, open-label, noninferior study to evaluate Acute Lumen Gain after dilatation. A total of 200 patients will be enrolled from 4 sites in China. All patients enrolled will be randomly assigned to the test group (DK ScoreTM group, n=100) and the control group (NSE group, n=100) with randomized allocation ratio of 1:1. Patients in the test group and the control group will be treated with DK ScoreTM Scoring balloon catheters or NSE Coronary Dilatation Catheter. A 30-day after procedure follow-up will be conducted for all 200 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients related

1. Age ≥ 18 years and ≤ 75 years.
2. Patients with symptomatic coronary artery disease with stable and unstable angina pectoralis remote myocardial infarction , asymptomatic subjects with coronary atherosclerotic stenosis causing myocardial ischemia.
3. Patients with indications for coronary artery bypass grafting.
4. Patients are able to follow protocol requirements and data collection procedures
5. Patients understand the purpose of the study, will voluntarily participate in the study and sign informed consent. Patients are willing to undergo clinical follow-up as required by this study.

Lesions Related:

1. Reference vessel diameter (RVD) between 2.0 and 4.0 mm by visual estimation.. Target lesion length ≤ 20 mm.
2. More than 70% stenosis (or more than 50% stenosis combined with symptoms of ischemia). TIMI≥1.
3. One target lesion needs to be Treated. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success as visually assessed by the physician. The non-target lesion need be located at another coronary artery different from the target lesion.
4. Investigator estimates that the target lesion need Cutting/Scoring balloon treatment. Target lesion is fully pre-dilated that scoring balloon is able to pass.

Exclusion Criteria:

Patients Related :

1. AMI within 1 week.
2. Patients has congestive heart failure or NYHA IV.
3. Renal dysfunctional (CRE>443umol/L).
4. Patient underwent heat transplant.
5. Pregnant or nursing.
6. Lifespan expectancy is less than 12 months
7. Patients with history of peptic ulcer or gastrointestinal bleeding, or the patients have a bleeding tendency evaluated by investigator. Patients are forbidden to use anticoagulation agents or anti-platelet drugs.
8. Patients are allergic to paclitaxel or heparin
9. Difficult for evaluation or treatment.
10. Patents are currently participating in another investigational drug or device study that has not yet completed its primary endpoint.
11. Patients participated in any other clinical trials less than 1 month.
12. Interventional surgery is expected to be extremely risky unsuitable for study evaluated by investigator.
13. Patient had poor compliance record and could not follow the study.

Lesion Related:

1. Target Lesion located in Left Main Artery lesions and Ostial lesion within 5mm to Left Main Artery.
2. Angiography shows thrombus in Target Lesion
3. Chronic Total Occlusion Lesion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Numerical Acute Lumen Gain in mm (QCA) | During the procedure
  Acute Lumen Gain for both arms will be measure with QCA, as accessed by independent core-lab.
  Angiographic endpoint will be in-lesion acute lumen gain defined as minimal lumen diameter (MLD) in lumen after dilatation by either arm device minus baseline MLD.

SECONDARY OUTCOMES:
Rate of Device success in percent | During the procedure
  Successful delivery to the target lesion, deployment, achieving less than 50% residual stenosis, and retrieval after procedure.
Rate of Target Lesion Failure in percent | 30±7 Days
  Defined as any Target Lesion Failure after procedure
Rate of Patient-oriented Composite Endpoint (POCE) in percent | 30±7 Days
  Patient-oriented Composite Endpoint after procedure
Rate of other Complications in percent | During the procedure
  Incidence of complications associated with the use of scoring balloon catheters
Rate of Clinical Success in percent | During the procedure
  Defined as <20% diameter stenosis after stenting for DCB, without in-hospital major adverse cardiac events/MI/TLR After PCI

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, Dr., Principal Investigator — Beijing Anzhen Hospital affiliated to Capital University of Medical
Locations (4):
- China (4):
  - Beijing Anzhen Hospital affiliated to Capital University of Medical, Beijing, Beijing Municipality
  - Xuzhou Third People Hospital, Xuzhou, Jiangsu
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Tianjin Chest Hospita, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No